CLINICAL TRIAL: NCT04877171
Title: Telemedicine Efficacy in Medication Adherence in Post-ischemic Stroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundación Cardiovascular de Colombia (Other)
Collaborators: Instituto Colombiano para el Desarrollo de la Ciencia y la Tecnología (COLCIENCIAS) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CEI-2020-01644
Record Dates: First submitted 2021-04-26; First posted 2021-05-07 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Stroke; Compliance, Patient; Compliance, Treatment; Compliance, Medication
Keywords: Stroke consultation; Telemedicine; Recovery; Rehabilitation
MeSH Terms: conditions — Stroke; Patient Compliance; Medication Adherence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- telemedicine neurology consultation (Experimental): Starting on day 12-14 post-discharge, participants will receive a phone call for a drug conciliation. Participants at 1-month post-discharge will receive a telemedicine consultation, another at 3 months and 6 months.
  Interventions: Other: telemedicine neurology consultation
- in-person neurology consultation (Active Comparator): Starting at 1-month post-discharge, participants will attend an in-person neurology consultation and the following consultations depend on their physician's criteria until completed 6 months post-discharge.
  Interventions: Other: in-person neurology consultation

INTERVENTIONS:
Other: telemedicine neurology consultation — consultations via phone-only at 12-14-day post-discharge. Consultations via phone both audio and video at 1, 3 and 6 months
  Arms: telemedicine neurology consultation
Other: in-person neurology consultation — consultation in-person at Hospital Internacional de Colombia
  Arms: in-person neurology consultation

SUMMARY:
Telemedicine is an incipient resource to support the stroke system of care in Colombia. Several studies had demonstrated that patients benefit by implementing telestroke, for instance, providing timely and appropriate neurological consultation, diminishing accessible barriers, improving medication adherence for secondary prevention and facilitating linkages between patient and physician, especially for those in rural or neurologically underserved areas.

Hypothesis: The use of Telemedicine improves medication adherence in Post-ischemic Stroke.

Study Design: This is a randomized, single-blind, clinical trial to assess the efficacy of Telemedicine, over medication adherence in Post-ischemic Stroke subjects from Colombia.

Population: Eighty-four Post-ischemic Stroke subjects, subjects of both genders, over 18 years old, with a first stroke will be included.

Ethical Aspects: The study will be conducted according to the Helsinki declaration, the good clinical practices guidelines and the Colombian legislation. Prior to entering the study, patients must sign a written or oral informed consent that has been approved by the Institutional Ethics Committee of Fundación Cardiovascular de Colombia.

Overall objective: this study aims to determine the efficacy of telemedicine on pharmacological adherence in post-ischemic Stroke Participants.

Focus of study: Adherence to secondary stroke prevention medication.

ELIGIBILITY:
Inclusion Criteria:

* First ischemic stroke.
* Lived in urban areas.
* Available Access to permanent internet at home, in work on mobile dispositive, computers or tablets.
* Patients who gave their written informed consent.

Exclusion Criteria:

* Diagnosis of neurodegenerative diseases such as dementia and Parkinson's disease.
* Diagnosis of Diseases-terminal to prevent tracking.
* Diagnosis of psychiatric illnesses such as major depressive disorder (MDD) or others.
* Global cognitive impairment or previous diagnosis of dementia.

Ages: 18 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2021-07-16 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-08-30 (Estimated)

PRIMARY OUTCOMES:
Percentage medication adherence through Morisky-Green questionnaire | 6 months
  The Morisky Medication Adherence Scale in the original version (MMAS-4) is a structured self-report measure of medication-taking behavior. It consists of 4 items, with binary scoring (yes/no). Patients score one point for every 'Yes' answer. A score of 0 indicates high adherence; a score of 1 or 2 indicates intermediate adherence, and a score of 3 or 4 indicates low adherence.

SECONDARY OUTCOMES:
The Fantastic lifestyle assessment questionnaire | 6 months
  The fantastic instrument consists of a questionnaire with 25 closed-end questions across nine domains of the physical, psychological, and social components of lifestyle. The 23 first questions have multiple-choice (five answers) and the last two are dichotomous. The sum of all points yields a total score that classifies individuals in five categories, as follows: "Excellent" (85 to 100 points), "Very good" (70 to 84 points), "Good" (55 to 69 points), "Regular" (35 to 54 points), and "Needing improvement" (0 to 34 points).
Caregiver burden questionnaire | 6 months
  The Zarit Burden instrument contains 22 items. Each item on the interview is a statement which the caregiver is asked to endorse using a 5-point scale. Response options range from 0 (Never) to 4 (Nearly Always) with the sum of scores ranging between 0-88. Higher scores are taken to indicate increased burden intensity (score: ≤21=no burden; 21-40 = mild burden; 41-60 = moderate burden; ≥61 = severe burden).

OTHER OUTCOMES:
Presence of adverse events related to secondary stroke prevention medication | 6 months
  Thirty days after beginning the treatment, and every consultation month thereafter, the participants will be asked about the occurrence of adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Internacional de Colombia, Piedecuesta, Santander Department, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Broderick JP, Abir M. Transitions of Care for Stroke Patients: Opportunities to Improve Outcomes. Circ Cardiovasc Qual Outcomes. 2015 Oct;8(6 Suppl 3):S190-2. doi: 10.1161/CIRCOUTCOMES.115.002288. No abstract available. PMID 26515208
- [Background] Kalanithi L, Tai W, Conley J, Platchek T, Zulman D, Milstein A. Better health, less spending: delivery innovation for ischemic cerebrovascular disease. Stroke. 2014 Oct;45(10):3105-11. doi: 10.1161/STROKEAHA.114.006236. Epub 2014 Aug 14. No abstract available. PMID 25123221
- [Background] Coleman EA, Parry C, Chalmers S, Min SJ. The care transitions intervention: results of a randomized controlled trial. Arch Intern Med. 2006 Sep 25;166(17):1822-8. doi: 10.1001/archinte.166.17.1822. PMID 17000937
- [Background] Naylor M, Brooten D, Jones R, Lavizzo-Mourey R, Mezey M, Pauly M. Comprehensive discharge planning for the hospitalized elderly. A randomized clinical trial. Ann Intern Med. 1994 Jun 15;120(12):999-1006. doi: 10.7326/0003-4819-120-12-199406150-00005. PMID 8185149
- [Background] Poston KM, Dumas BP, Edlund BJ. Outcomes of a quality improvement project implementing stroke discharge advocacy to reduce 30-day readmission rates. J Nurs Care Qual. 2014 Jul-Sep;29(3):237-44. doi: 10.1097/NCQ.0000000000000040. PMID 24322371
- [Background] Ogren J, Irewall AL, Soderstrom L, Mooe T. Long-term, telephone-based follow-up after stroke and TIA improves risk factors: 36-month results from the randomized controlled NAILED stroke risk factor trial. BMC Neurol. 2018 Sep 21;18(1):153. doi: 10.1186/s12883-018-1158-5. PMID 30241499
- [Background] Cameron JI, O'Connell C, Foley N, Salter K, Booth R, Boyle R, Cheung D, Cooper N, Corriveau H, Dowlatshahi D, Dulude A, Flaherty P, Glasser E, Gubitz G, Hebert D, Holzmann J, Hurteau P, Lamy E, LeClaire S, McMillan T, Murray J, Scarfone D, Smith EE, Shum V, Taylor K, Taylor T, Yanchula C, Teasell R, Lindsay P; Heart and Stroke Foundation Canadian Stroke Best Practice Committees. Canadian Stroke Best Practice Recommendations: Managing transitions of care following Stroke, Guidelines Update 2016. Int J Stroke. 2016 Oct;11(7):807-22. doi: 10.1177/1747493016660102. Epub 2016 Jul 21. PMID 27443991
- [Background] Duncan PW, Bushnell CD, Rosamond WD, Jones Berkeley SB, Gesell SB, D'Agostino RB Jr, Ambrosius WT, Barton-Percival B, Bettger JP, Coleman SW, Cummings DM, Freburger JK, Halladay J, Johnson AM, Kucharska-Newton AM, Lundy-Lamm G, Lutz BJ, Mettam LH, Pastva AM, Sissine ME, Vetter B. The Comprehensive Post-Acute Stroke Services (COMPASS) study: design and methods for a cluster-randomized pragmatic trial. BMC Neurol. 2017 Jul 17;17(1):133. doi: 10.1186/s12883-017-0907-1. PMID 28716014
- [Background] Ross L, Bena J, Bermel R, McCarter L, Ahmed Z, Goforth H, Cherian N, Kriegler J, Estemalik E, Stanton M, Rasmussen P, Fernandez HH, Najm I, McGinley M. Implementation and Patient Experience of Outpatient Teleneurology. Telemed J E Health. 2021 Mar;27(3):323-329. doi: 10.1089/tmj.2020.0032. Epub 2020 Jun 23. PMID 32584654
- [Background] Appireddy R, Khan S, Leaver C, Martin C, Jin A, Durafourt BA, Archer SL. Home Virtual Visits for Outpatient Follow-Up Stroke Care: Cross-Sectional Study. J Med Internet Res. 2019 Oct 7;21(10):e13734. doi: 10.2196/13734. PMID 31593536
- [Background] Morisky DE, Green LW, Levine DM. Concurrent and predictive validity of a self-reported measure of medication adherence. Med Care. 1986 Jan;24(1):67-74. doi: 10.1097/00005650-198601000-00007. PMID 3945130
- [Background] Zarit SH, Reever KE, Bach-Peterson J. Relatives of the impaired elderly: correlates of feelings of burden. Gerontologist. 1980 Dec;20(6):649-55. doi: 10.1093/geront/20.6.649. No abstract available. PMID 7203086